CLINICAL TRIAL: NCT02817035
Title: Study of Neural Inspiratory Time and Expiratory Delay in Patients and Healthy Subjects During Unassisted Spontaneous Breathing and Mechanical Ventilation.
Brief Title: Study of Neural Inspiratory Time and Expiratory Delay in Patient and Health During Spontaneous Breathing and Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhang Jianheng, Dr, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: yls2016
Record Dates: First submitted 2016-06-16; First posted 2016-06-29 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: State Key Laboratory of Respiratory Disease
Keywords: interstitial lung disease; chronic obstructive pulmonary disease; mechanical ventilation; expiratory delay; neural inspiratory time
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- noninvasive mechanical ventilation (Experimental): To investigate the change of the neural inspiratory time and expiratory delay noninvasive mechanical ventilation ,in comparison to spontaneous breathing
  Interventions: Device: noninvasive mechanical ventilation

INTERVENTIONS:
Device: noninvasive mechanical ventilation — To examined the physiological signals of patients and healthy subjects during spontaneous breathing and noninvasive mechanical ventilation.

SUMMARY:
To make these definitions of neural inspiratory time (Ti) and expiratory delay clearly.The present study was undertaken to examined the physiological signals of patients and healthy subjects during spontaneous breathing and noninvasive mechanical ventilation.

DETAILED DESCRIPTION:
In total, 8 chronic obstructive pulmonary disease (COPD) patients, 8 patients with interstitial lung disease (ILD) and 8 healthy subjects were recruited.

The patient was studied at the afternoon in a semirecumbent position. After the application of topical anaesthesia (2% xylocaine), the patient was asked to swallow two balloon-tipped catheters and the multi-pair esophageal electrode catheter through the nose into the their right position.

At the first period, the stable signals of unassisted spontaneous breathing (about 5min) were chosen to be recorded. After this period, the patient was placed on noninvasive pressure support ventilation(PSV). The inspiratory positive airway pressure (IPAP) was initially titrated by patient's tolerance . The noninvasive ventilation lasted at least 20 minutes until the breathing was stable. All the raw signals were recorded. The last 15 minutes of the stable computer-stored data were calculated and analyzed. The leaks were monitored by the display of the ventilator and the computer during the procedure. When the leak was observed, the mask was carefully adjusted to prevent. Esophageal and gastric balloon-catheters were used to detect the intra-thoracic and abdominal pressure. Airway pressure was also measured simultaneously. EMGdi was recorded from a multipair esophageal electrode .During ventilation Airflow and ventilation were measured with pneumotachograph.

Respiratory rate, tidal volume,the time difference between the initial increase and the termination of the diaphragm electromyogram(EMGdi) , time difference between maximal value of EMGdi and the end of inspiratory flow,time difference between the point of zero flow between inspiration and expiration ,and the time difference between the onset of the upward deflection in transdiagramic pressure( Pdi) and the return of Pdi were calculated during the unassisted spontaneous breathing and mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. chronic obstructive pulmonary disease patient meet the diagnose criteria of chronic obstructive pulmonary disease
2. interstitial lung disease patient meet the diagnose criteria of interstitial lung disease
3. healthy subjects No history of the lung and Cardiovascular disease.The lung function is normal.

Exclusion Criteria:

1. severe Cardiovascular disease
2. Pneumonia
3. neuromuscular and chest wall deformity
4. Respiratory arrest
5. Cardiovascular instability (hypotension, arrhythmias, myocardial infarction)
6. Change in mental status; uncooperative patient
7. High aspiration risk
8. Viscous or copious secretions
9. Recent facial or gastroesophageal surgery
10. Craniofacial trauma
11. Fixed nasopharyngeal abnormalities
12. Burns
13. Extreme obesity

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
neural inspiratory time | 20-30 minutes
  Compare the neural inspiratory time during spontaneous breathing and noninvasive mechanical ventilation.

SECONDARY OUTCOMES:
expiratory delay | 20-30 minutes
  to assess the expiratory delay during noninvasive mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: rongchang chen, MD, Study Director — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- TheFirst Affiliated Hospital Of Guangzhou Medical Collage, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided